CLINICAL TRIAL: NCT06397365
Title: Effect of Hypnosis on Adherence to Continuous Positive Airway Pressure Therapy in Sleep-disordered Breathing: a Randomized Controlled Trial
Brief Title: Effect of Hypnosis on Adherence to Continuous Positive Airway Pressure.
Acronym: HypnOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solelhac Geoffroy (Other)
Responsible Party: Sponsor-Investigator, Solelhac Geoffroy, MD, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUVaudois-HypnOSA
Record Dates: First submitted 2024-04-23; First posted 2024-05-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Apnea Syndrome; Apnea, Obstructive
Keywords: CPAP adherence; medical hypnosis; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypnosis (Experimental): Baseline study visit (V1): signature of the informed consent form, verification of eligibility criteria, collection of demographic data, polygraphy or polysomnography features, data provided by the CPAP machine (one month), questionnaires.
  During the second visit (V2), the patient randomized in HYP group will come for the hypnosis sessions.
  Follow-up visit (V4): 28-42 days (4-6 weeks) after V3 for HYP group and 2 months (+/- 14 days) after V1 for SOC group. Collection of data provided by the CPAP machine (one month), questionnaires.
  Interventions: Other: medical hypnosis
- standard of care (No Intervention): Baseline study visit (V1): signature of the informed consent form, verification of eligibility criteria, collection of demographic data, polygraphy or polysomnography features, data provided by the CPAP machine (one month), questionnaires.
  Usual management of CPAP treatment by the home care provider and the prescribing doctor without any change in management.
  Follow-up visit (V4): 28-42 days (4-6 weeks) after V3 for HYP group and 2 months (+/- 14 days) after V1 for SOC group. Collection of data provided by the CPAP machine (one month), questionnaires.

INTERVENTIONS:
Other: medical hypnosis — The first hypnosis session (V2) consists of a safe place suggestion. Through this type of suggestions, patients will safely experience the dissociative state, and will be given tools (recordings of sessions) to perform self-hypnosis at home between the visits. The suggestions will help the patient to visualize an imaginary place where they feel well and safe, a protective place to rest. In this first session, CPAP treatment will be introduced during hypnosis, with specific suggestions relating to the use of this treatment.
  The second session (V3) The second session will also use the safe place. We will adapt the suggestions according to the experience reported by the patient on the day of the visit. During this session, we'll focus on changes in the patient's perception of the CPAP machine.
  Patients will also be given the recording of each session to perform self-hypnosis at home between the visits.
  Arms: Hypnosis

SUMMARY:
The prevalence of sleep-disordered breathing is high, with an apnea-hypopnea index of over 15 per hour found in 49.7% of men and 23.4% of women in the general population (1). The gold standard treatment for sleep-disordered breathing is continuous positive airway pressure (CPAP) therapy (2). However, nearly 30% of patients are considered non-adherent to CPAP treatment (3). Moreover, the number of hours of CPAP usage has been shown to be directly associated with a reduction in objective and subjective sleepiness, and improvement in daytime functioning (4). A recent prospective study conducted in a French clinical population cohort of 5138 participants found an effect of CPAP treatment duration on reducing the risk of developing a major cardiovascular event (stroke, myocardial infarction, all-cause mortality) (5). Therefore, the poor adherence to CPAP treatment represents a public health challenge for healthcare professionals managing these patients. Several predictors for non-adherence can be identified, such as using CPAP for less than 4 hours per night during the initial treatment phase, moderate to severe obstructive sleep apnea, or low self-esteem (6). Measures aimed at promoting patient adaptation from the initiation of treatment are crucial as this period determines long-term adherence to CPAP therapy (7). Among these measures, there is the management of "physical" adverse effects such as xerostomia (using a humidifier), feeling too much or too little air (modifying CPAP pressure profiles), skin problems, and mask air leaks (interface adjustment), which are well-known and applied by health care organization providing the CPAP machines (2).

On top of these "technical" problems, patients related issues such as mask-induced anxiety, psychosocial conditions, and dysfunctional thoughts about CPAP treatment may prevent patients from using their CPAP properly. Innovative tools such as psycho corporal therapies, including medical hypnosis, could be used in these situations. A recent literature review focusing on the impact of medical hypnosis on sleep disorders in adult patients found an improvement in various sleep parameters (sleep quality, insomnia complaints, frequency and/or intensity of parasomnias) in 58.4% of patients. However, in this systematic review of 24 studies, none of them explored the use of medical hypnosis in sleep-related breathing disorders (8).

Hypnosis can be defined as an altered state of consciousness in which a person's attention is detached from their immediate environment and absorbed in inner experiences such as feelings, cognition, and imagery (9). Hypnotic induction involves focusing attention and imaginative involvement to the point where what is imagined seems real. By using and accepting suggestions, the clinician and the patient create a benevolent hypnotic reality with the goal of improving the patient's clinical situation (10).

In the literature, there is only one clinical case report describing a benefit of medical hypnosis for CPAP tolerance in a child with cherubism (a rare fibro-osseous genetic disease-causing nasal obstruction). In this case, CPAP therapy using an oral interface was fully accepted after three hypnosis sessions and corrected the obstructive sleep breathing disorder (11). In a slightly different domain, there is a case report of successful use of medical hypnosis as an adjunct therapy for weaning from mechanical ventilation (12).

Our hypothesis is that the use of medical hypnosis in CPAP-treated patients could improve the patient's perception of the treatment, making it more positive. Medical hypnosis could occur very early in the management process, with rapid learning of self-hypnosis to actively influence this crucial period for long term adherence of CPAP. The principal objective is therefore to evaluate the effects of medical hypnosis on adherence to CPAP therapy in patients with sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Indication for long-term CPAP treatment for sleep-disordered breathing.
* Intolerance of CPAP with use of less than 3h/night on average (assessed at the second CPAP check-up by the home care provider 1 to 3 months CPAP introduction).
* Ability to provide informed consent.

Exclusion Criteria:

* Patient's refusal to experience hypnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
average hours of CPAP | Baseline after randomisation and at last visit 6 weeks after randomisation
  average hours of CPAP use before and after the hypnosis therapy.

SECONDARY OUTCOMES:
nights with CPAP use of more than 4 hours | Baseline after randomisation and at last visit 6 weeks after randomisation
  percentage of nights with CPAP use of more than 4 hours before and after the hypnosis therapy
patients continuing to use CPAP | Baseline after randomisation and at last visit 6 weeks after randomisation
  percentage of patients continuing to use CPAP at the end of the study.
sleepiness | Baseline after randomisation and at last visit 6 weeks after randomisation
  Epworth Sleepiness Scale to evaluate daytime sleepiness. (0 to 24. The higher the score, the higher that person's average sleep propensity in daily life or their daytime sleepiness)
sleep quality | Baseline after randomisation and at last visit 6 weeks after randomisation
  Pittsburgh Sleep Quality Index to evaluate sleep quality over a 1-month period. (0 to 21 points, where 0 means that there are no difficulties, and 21 indicating major difficulties.)
Insomnia | Baseline after randomisation and at last visit 6 weeks after randomisation
  Evaluation of the diagnosis of chronic insomnia according to the Insomnia Severity Index.(0 to 28 :
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe))
Score at the Quebec Sleep Questionnaire | Baseline after randomisation and at last visit 6 weeks after randomisation
  Quebec Sleep Questionnaire to evaluate the quality of life related specifically to obstructive sleep apnea. The questionnaire assesses five domains: (1) hypersomnolence; (2) diurnal symptoms; (3) nocturnal symptoms; (4) emotions; and (5) social interactions. Each domain includes 4-7 items and each item is scored on a 7-point scale. For each domain, higher scores indicates milder symptoms.
Anxiety and emotion | Baseline after randomisation and at last visit 6 weeks after randomisation
  The Hospital Anxiety and Depression Scale to evaluate the psychological state. The scale is an instrument for screening for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety and seven others to the depressive dimension. two scores (maximum score for each = 21). A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUVaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No